CLINICAL TRIAL: NCT05581199
Title: A Phase 2b, Multi-center, Randomized, Quadruple-blind, Placebo-controlled Study of Batoclimab Treatment in Adult Participants With Active Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: To Assess Efficacy and Safety of Batoclimab in Adult Participants With Active CIDP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMVT-1401-2401
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Chronic Inflammatory Demyelinating Polyneuropathy; IMVT-1401; Monoclonal antibody; Autoimmune disorders
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Autoimmune Diseases | interventions — Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Treatment Period 1: Cohort A, Dose 1 (Experimental)
  Interventions: Drug: Batoclimab 680 milligrams (mg) subcutaneous (SC) weekly
- Treatment Period 1: Cohort A, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Treatment Period 1: Cohort B, Dose 1 (Experimental)
  Interventions: Drug: Batoclimab 680 milligrams (mg) subcutaneous (SC) weekly
- Treatment Period 1: Cohort B, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Treatment Period 1: Cohort C, Dose 1 (Experimental)
  Interventions: Drug: Batoclimab 680 milligrams (mg) subcutaneous (SC) weekly
- Treatment Period 1: Cohort C, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Treatment Period 1: Cohort D, Dose 1 (Experimental)
  Interventions: Drug: Batoclimab 680 milligrams (mg) subcutaneous (SC) weekly
- Treatment Period 1: Cohort D, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Withdrawal Period 2: Cohort A, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Withdrawal Period 2: Cohort A, Placebo (Experimental)
  Interventions: Drug: Placebo
- Withdrawal Period 2: Cohort B, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Withdrawal Period 2: Cohort B, Placebo (Experimental)
  Interventions: Drug: Placebo
- Withdrawal Period 2: Cohort C, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Withdrawal Period 2: Cohort C, Placebo (Experimental)
  Interventions: Drug: Placebo
- Withdrawal Period 2: Cohort D, Dose 2 (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Withdrawal Period 2: Cohort D, Placebo (Experimental)
  Interventions: Drug: Placebo
- LTE Period: With Relapse in Period 2: Dose 1 and Dose 2 (Experimental): Participants will receive Dose 1 for the initial 4 weeks only and Dose 2 for the remaining 48 weeks.
  Interventions: Drug: Batoclimab 680 milligrams (mg) subcutaneous (SC) weekly; Drug: Batoclimab 340 mg SC weekly
- LTE Period: Without Relapse in Period 2: Dose 2 (Experimental): Participants will receive Dose 2 for all 52 weeks.
  Interventions: Drug: Batoclimab 340 mg SC weekly

INTERVENTIONS:
Drug: Batoclimab 680 milligrams (mg) subcutaneous (SC) weekly — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody
  Other Names: IMVT-1401
  Arms: LTE Period: With Relapse in Period 2: Dose 1 and Dose 2; Treatment Period 1: Cohort A, Dose 1; Treatment Period 1: Cohort B, Dose 1; Treatment Period 1: Cohort C, Dose 1; Treatment Period 1: Cohort D, Dose 1
Drug: Batoclimab 340 mg SC weekly — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody
  Other Names: IMVT-1401
  Arms: LTE Period: With Relapse in Period 2: Dose 1 and Dose 2; LTE Period: Without Relapse in Period 2: Dose 2; Treatment Period 1: Cohort A, Dose 2; Treatment Period 1: Cohort B, Dose 2; Treatment Period 1: Cohort C, Dose 2; Treatment Period 1: Cohort D, Dose 2; Withdrawal Period 2: Cohort A, Dose 2; Withdrawal Period 2: Cohort B, Dose 2; Withdrawal Period 2: Cohort C, Dose 2; Withdrawal Period 2: Cohort D, Dose 2
Drug: Placebo — Matching placebo SC
  Arms: Withdrawal Period 2: Cohort A, Placebo; Withdrawal Period 2: Cohort B, Placebo; Withdrawal Period 2: Cohort C, Placebo; Withdrawal Period 2: Cohort D, Placebo

SUMMARY:
This is a multi-center, randomized, quadruple-blind, placebo-controlled study to evaluate the efficacy and safety of batoclimab in adult participants with active CIDP. The study includes an up to 4-week Screening Period, an up to 12-week Washout Period, a 12-week Randomized Treatment Period (Period 1), an up to 24-week Randomized Withdrawal Period (Period 2), an up to 52-week Long-term Extension (LTE) Period (optional), and Safety Follow-up 4 weeks after the last dose of study treatment. The total study duration will be up to approximately 109 weeks. Eligible participants will be assigned to one of four cohorts based upon their baseline CIDP treatment (Cohorts A and D - immunoglobulin [Ig] or plasma exchange [PLEX]; Cohort B - corticosteroids; Cohort C - naive or untreated in previous 3-24 months) and whether they meet diagnosis according to the European Academy of Neurology/Peripheral Nerve Society (EAN/PNS) criteria (Cohorts A, B, and C) or clinical criteria only (Cohort D) at the time of screening.

ELIGIBILITY:
Inclusion criteria:

All Cohorts:

1. Are >= 18 years at the Screening Visit.
2. Have met clinical diagnostic criteria for typical CIDP, or one of the following CIDP variants: multifocal CIDP, focal CIDP, or motor CIDP in accordance with the EAN/PNS Guideline on Diagnosis and Treatment of CIDP. Clinical criteria for typical CIDP and variants are as follows (either criterion must be met):

   1. Typical CIDP: All the following:

      * Progressive or relapsing, symmetric, proximal, and distal muscle weakness of upper and lower limbs, and sensory involvement of at least two limbs (at any point in the disease course)
      * Developing over at least 8 weeks
      * Absent or reduced tendon reflexes in all limbs
   2. CIDP variants: One of the following, but otherwise as in typical CIDP (tendon reflexes may be normal in unaffected limbs):

      * Multifocal CIDP: documented sensory loss and muscle weakness in a multifocal pattern, usually asymmetric, upper limb predominant
      * Focal CIDP: sensory loss and muscle weakness in only one limb
      * Motor CIDP: motor symptoms and signs without sensory involvement

   Cohorts A and B:
3. Have electrodiagnostic test results supporting the diagnosis of CIDP in accordance with the EAN/PNS Guideline on Diagnosis and Treatment of CIDP; for Cohorts A and B, either criterion must be met:

   1. Motor nerve conduction criteria strongly supportive of demyelination.
   2. Motor nerve conduction criteria weakly supportive of demyelination and 2 or more of the following additional diagnostic criteria:

      * Objective improvement to an empiric trial of therapy with immunoglobulin treatment, plasma exchange (PLEX), or corticosteroids.
      * Diagnostic imaging by ultrasound or magnetic resonance imaging (MRI) supporting the diagnosis of CIDP by demonstrating nerve enlargement.
      * Cerebrospinal fluid (CSF) demonstrating albuminocytologic dissociation (i.e., elevated CSF protein level [defined as > 70 milligrams per deciliter {mg/dL} or > 10 mg/dL greater than years of age for those aged 60 years and over] with normal CSF white blood cell [WBC] level).
      * Nerve biopsy demonstrating features supporting the diagnosis of CIDP, such as edema, demyelination, and/or onion bulb formation.

   Cohort C only:
4. Have a diagnosis of CIDP in accordance with the EAN/PNS Guideline on Diagnosis and Treatment of CIDP based on clinical criteria and motor nerve conduction criteria strongly supportive of demyelination (i.e., motor nerve conduction criteria weakly supportive of demyelination is insufficient diagnostic evidence for admission to Cohort C).

   Cohort D only:
5. Have met only clinical diagnostic criteria for typical CIDP, or one of the following CIDP variants: multifocal CIDP, focal CIDP, or motor CIDP in accordance with the EAN/PNS Guideline on Diagnosis and Treatment of CIDP. Either inclusion criterion 2(a) or 2(b) must be met.

Additional inclusion criteria are defined in the protocol.

Exclusion Criteria:

All Cohorts:

1. Have current or prior history of immunoglobulin M (IgM) paraproteinemia with or without anti-myelin-associated-glycoprotein antibodies.
2. Have Distal CIDP, Sensory CIDP or are suspected of having a diagnosis of auto-immune nodopathy in accordance with the EAN/PNS Guideline on Diagnosis and Treatment of CIDP.
3. Have polyneuropathy of causes other than CIDP including but not limited to:

   1. Multifocal motor neuropathy
   2. Hereditary demyelinating neuropathy
   3. Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin change syndromes (i.e., POEMS)
   4. Lumbosacral radiculoplexus neuropathy
   5. Systemic illnesses including vitamin deficiency syndromes and paraneoplastic neuropathies
   6. Drug- or toxin-induced
4. Have diabetes mellitus (DM) and meets any of the following criteria:

   1. Does not meet inclusion criteria 2(a) and 3(a).
   2. In the opinion of the Investigator, there is evidence of poorly controlled DM preceding the diagnosis of CIDP.
   3. In the opinion of the Investigator, there is evidence of poorly controlled DM at screening.
5. Have a history of myelopathy or evidence of central demyelination.
6. Are receiving chronic oral corticosteroids monotherapy at a dose > 40 mg/day prednisolone/prednisone or its equivalent at the Screening Visit.
7. Are receiving chronic oral corticosteroid at a dose > 10 mg/day prednisolone/prednisone or equivalent in combination with immunoglobulin therapy or PLEX at the Screening Visit.

Additional exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Period 2, Cohort A: Proportion of participants who remain relapse-free at Week 36 | Week 36
  Relapse is defined as a worsening (increase) of >=1 point on adjusted inflammatory neuropathy cause and treatment (AdjINCAT) score at any time point during Period 2 relative to Period 2 Baseline which is sustained at a Follow-Up visit 1 week later. The INCAT disability scale is a widely used and validated efficacy assessment of neurologic dysfunction in CIDP. Upper and lower limb dysfunction are each separately assessed on a scale of 0-5 and results are summed together for a total composite score of 0-10. Higher scores represent greater disability. The Adj INCAT disability score is identical to INCAT disability score with exception that changes in upper limb function from 0 (normal) to 1 (minor symptoms) and vice versa are excluded since minor symptoms in the fingers, which are implied by an upper limb score of 1, are not considered clinically significant in all participants. The Adj INCAT disability score will be used for participant selection and measurement of clinical response.

SECONDARY OUTCOMES:
Period 2, Cohort A: Time to first relapse relative to Period 2 Baseline | Baseline (Week 12) to Week 36
Period 2, Cohort A: Change from Period 2 Baseline in Adj INCAT score | Baseline (Week 12) and up to Week 36
Period 2, Cohort A: Change from Period 2 Baseline in Inflammatory Rasch-built Overall Disability Scale (I-RODS) | Baseline (Week 12) and up to Week 36
  The I-RODS for immune-mediated peripheral neuropathies is a patient-based linearly weighted scale that captures activity and social participation limitations in patients with CIDP. The assessment consists of a 24-question instrument that addresses upper and lower limb tasks that range in difficulty from reading a book and eating to standing and running. Answers are scored on a scale of 0-2 (complete disability to no disability) and the raw scores are then transformed into a final score ranging from 0-100.
Period 2, Cohort A: Change from Period 2 Baseline in Mean grip strength | Baseline (Week 12) and up to Week 36
  Mean Grip strength provides an objective, quantitative and immediate assessment of strength impairment. The Jamar dynamometer and the Martin vigorimeter are both commonly used to assess mean grip strength.
Period 2, Cohort A: Change from Period 2 Baseline in Medical Research Council (MRC) Sum Score | Baseline (Week 12) and up to Week 36
  The MRC sum score is a standardized methodology for objectively assessing and reporting muscle function. Six muscle groups are assessed bilaterally, and each scored on a scale of 0 (no visible contraction) to 5 (normal) yielding a sum ranging from 0 (paralysis) to 60 (normal strength). Higher scores indicate normal muscle strength.
Period 2, Cohort A: Change from Period 2 Baseline in Overall Neuropathy Limitations Scale (ONLS) | Baseline (Week 12) and up to Week 36
  The ONLS is a scale that focuses on upper and lower limb functions and was designed to assess the limitations of participants with immune-mediated peripheral neuropathies. This scale is completed by adding the total of the arm grade from zero point (less limitation) to 5 points (most limitation) and leg grade from zero point (less limitation) to 7 points (more limitation) yielding a total score of 0 (no disability) to 12 (maximum disability). Lower values in the ONLS indicate a better clinical condition.
Period 2, Cohorts A and B combined: Change from Period 2 Baseline in Adj INCAT score | Baseline (Week 12) and up to Week 36
Period 2, Cohorts A and B combined: Change from Period 2 Baseline in I-RODS | Baseline (Week 12) and up to Week 36
Period 2, Cohorts A and B combined: Change from Period 2 Baseline in Mean Grip Strength | Baseline (Week 12) and up to Week 36
Period 2, Cohorts A and B combined: Change from Period 2 Baseline in MRC sum score | Baseline (Week 12) and up to Week 36
Period 2, Cohorts A and B combined: Change from Period 2 Baseline in ONLS | Baseline (Week 12) and up to Week 36
Period 2, Cohorts A, B, and C: Proportion of participants who remain relapse-free at Week 36 | Week 36

CONTACTS AND LOCATIONS:
Locations (116):
- United States (33):
  - Site Number - 1603, Scottsdale, Arizona
  - Site Number - 1618, Carlsbad, California
  - Site Number - 1634, Los Angeles, California
  - Site Number - 1619, Orange, California
  - Site Number - 1608, San Francisco, California
  - Site Number - 1625, Aurora, Colorado
  - Site Number - 1636, Fort Collins, Colorado
  - Site Number - 1621, New Haven, Connecticut
  - Site Number - 1630, Washington D.C., District of Columbia
  - Site Number - 1600, Boca Raton, Florida
  - Site Number - 1609, Jacksonville, Florida
  - Site Number - 1631, Orlando, Florida
  - Site Number - 1629, Orlando, Florida
  - Site Number - 1617, Ormond Beach, Florida
  - Site Number - 1620, Port Charlotte, Florida
  - Site Number - 1633, Rockledge, Florida
  - Site Number - 1604, St. Petersburg, Florida
  - Site Number - 1607, O'Fallon, Illinois
  - Site Number - 1602, Kansas City, Kansas
  - Site Number - 1611, Nicholasville, Kentucky
  - Site Number - 1622, Brooklyn, New York
  - Site Number - 1605, New York, New York
  - Site Number - 1635, Chapel Hill, North Carolina
  - Site Number - 1610, Charlotte, North Carolina
  - Site Number - 1614, Portland, Oregon
  - Site Number - 1623, Philadelphia, Pennsylvania
  - Site Number - 1624, Philadelphia, Pennsylvania
  - Site Number -1601, Austin, Texas
  - Site Number - 1606, Houston, Texas
  - Site Number - 1628, San Antonio, Texas
  - Site Number - 1627, Richmond, Virginia
  - Site Number - 1632, Seattle, Washington
  - Site Number - 1613, Milwaukee, Wisconsin
- Argentina (4):
  - Site Number - 7753, Rosario, Santa Fe Province
  - Site Number - 7751, Rosario, Santa Fe Province
  - Site Number - 7752, San Miguel de Tucumán, Tucumán Province
  - Site Number - 7750, Buenos Aires
- Belgium (2):
  - Site Number - 4681, Ghent, Oost-Vlaanderen
  - Site Number - 4680, Leuven, Vlaams Brabant
- Brazil (5):
  - Site Number - 9103, Brasília, Federal District
  - Site Number - 9101, Curitiba, Paraná
  - Site Number - 9100, Ribeirão Preto, São Paulo
  - Site Number - 9102, Rio de Janeiro
  - Site Number - 9105, São Paulo
- Bulgaria (3):
  - Site Number - 9111, Sofia, Sofia-Grad
  - Site Number - 9110, Sofia, Sofia-Grad
  - Site Number - 9112, Pleven
- Canada (2):
  - Site Number - 2600, Edmonton, Alberta
  - Site Number - 2603, Vancouver, British Columbia
- Site Number - 4740, Copenhagen, Denmark
- Site Number - 3241, Turku, Southwest Finland, Finland
- Germany (5):
  - Site Number - 6704, München, Bavaria
  - Site Number - 6705, Bochum, North Rhine-Westphalia
  - Site Number - 6700, Dresden, Saxony
  - Site Number - 6702, Leipzig, Saxony
  - Site Number - 6706, Berlin
- Greece (7):
  - Site Number - 6341, Pátrai, Achaïa
  - Site Number - 6344, Athens, Attica
  - Site Number - 6345, Athens, Attica
  - Site Number - 6343, Alexandroupoli, Evros
  - Site Number - 6346, Ioannina, Ioannina
  - Site Number - 6342, Heraklion, Irakleio
  - Site Number - 6347, Larissa
- Italy (10):
  - Site Number - 6302, Gussago, Brescia
  - Site Number - 6305, Bologna, Emilia-Romagna
  - Site Number - 6304, Udine, Friuli Venezia Giulia
  - Site Number - 6309, Rome, Lazio
  - Site Number - 6306, Rome, Lazio
  - Site Number - 6301, Bergamo, Lombardy
  - Site Number - 6307, Milan, Lombardy
  - Site Number - 6303, Pisa, Tuscany
  - Site Number - 6308, Siena, Tuscany
  - Site Number - 6300, Pavia
- Site Number - 6491, Oslo, Norway
- Poland (12):
  - Site Number - 3207, Poznan, Greater Poland Voivodeship
  - Site Number - 3211, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Site Number - 3203, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Site Number - 3208, Krakow, Lesser Poland Voivodeship
  - Site Number - 3209, Krakow, Lesser Poland Voivodeship
  - Site Number - 3200, Krakow, Lesser Poland Voivodeship
  - Site Number - 3204, Wroclaw, Lower Silesian Voivodeship
  - Site Number - 3210, Lublin, Lublin Voivodeship
  - Site Number - 3206, Lublin, Lublin Voivodeship
  - Site Number - 3202, Mazurki, Lublin Voivodeship
  - Site Number - 3205, Gdansk, Pomeranian Voivodeship
  - Site Number - 3201, Katowice, Silesian Voivodeship
- Portugal (5):
  - Site Number - 3742, Senhora da Hora, Porto District
  - Site Number - 3745, Vila Nova de Gaia, Porto District
  - Site Number - 3743, Almada, Setúbal District
  - Site Number - 3741, Lisbon
  - Site Number - 3744, Porto
- Romania (4):
  - Site Number - 8406, Bucharest, București
  - Site Number - 8401, Târgu Mureş, Mureș County
  - Site Number - 8403, Timișoara, Timiș County
  - SIte Number - 8400, Constanța
- Serbia (4):
  - Site Number - 8501, Belgrade
  - Site Number - 8502, Belgrade
  - Site Number - 8500, Niš
  - Site Number - 8503, Novi Sad
- Slovakia (4):
  - Site Number - 8600, Liptovský Mikuláš
  - Site Number - 8601, Martin
  - Site Number - 8603, Prešov
  - Site Number - 8602, Trnava
- South Korea (2):
  - Site Number - 9901, Seoul
  - Site Number - 9900, Seoul
- Spain (4):
  - Site Number - 3701, L'Hospitalet de Llobregat, Barcelona
  - Site Number - 3704, Sant Cugat del Vallès, Barcelona
  - Site Number - 3700, San Sebastián, Gipuzkoa
  - Site Number - 3703, Barcelona
- Site Number - 4891, Gothenburg, Västra Götaland County, Sweden
- United Kingdom (6):
  - Site Number - 7405, Cambridge, Cambridgeshire
  - Site Number - 7402, Southampton, Hampshire
  - Site Number - 7404, Glasgow, Lanarkshire
  - Site Number - 7403, Preston, Lancashire
  - Site Number - 7401, Sheffield, South Yorkshire
  - Site Number - 7400, Manchester

IPD SHARING:
Plan to Share IPD: No